CLINICAL TRIAL: NCT02400905
Title: MIMICS-2: Evaluation of Safety and Effectiveness of the BioMimics 3D Stent System in the Femoropopliteal Arteries of Patients With Symptomatic Peripheral Arterial Disease
Brief Title: Evaluation of Safety and Effectiveness of the BioMimics 3D Stent System
Acronym: MIMICS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veryan Medical Ltd. (Industry)
Collaborators: ClinLogix. LLC (Industry); Yale Cardiovascular Research Group (Other); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CID-100
Record Dates: First submitted 2015-03-23; First posted 2015-03-27 (Estimated); Results first posted 2019-01-18 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; PVD; SFA stent
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BioMimics 3D Vascular Stent (Experimental): Implantation of BioMimics 3D nitinol stent using the BioMimics 3D Vascular Stent System
  Interventions: Device: BioMimics 3D Vascular Stent System

INTERVENTIONS:
Device: BioMimics 3D Vascular Stent System — Femoropopliteal stenting

SUMMARY:
To demonstrate that the BioMimics 3D Stent System meets the performance goals defined by VIVA Physicians, Inc. for the safety and effectiveness of Nitinol stents used in the treatment of symptomatic disease of the femoropopliteal artery. It is a prospective, single-arm, multicenter clinical trial.

DETAILED DESCRIPTION:
The BioMimics 3D stent is intended to improve luminal diameter in the treatment of symptomatic de-novo, obstructive or occlusive lesions in native femoropopliteal arteries with reference vessel diameters ranging from 4.0 - 6.0 mm. Subjects with symptomatic atherosclerotic disease of the femoropopliteal artery who comply with all study eligibility criteria may be considered for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic peripheral arterial disease (PAD) of the lower extremities requiring intervention to relieve de novo obstruction or occlusion of the native femoropopliteal artery.
* PAD classified as Rutherford clinical category 2, 3 or 4.
* Resting ankle-brachial index (ABI) of ≤0.90 (or ≤0.75 after exercise of the target limb) or angiographic or DUS evidence of >/= 60%.
* Single or multiple stenotic or occlusive lesions within the native femoropopliteal artery ("target lesions") that can be crossed with a guidewire and fully dilated.
* Single or multiple target lesions must be covered by a single stent or two overlapping stents.
* Target lesion(s) eligible for treatment at least 1 cm distal to the origin of the deep femoral artery and at least 3 cm above the bottom of the femur.
* Target lesion(s) reference vessel diameter is between 4.0 mm and 6.0 mm.
* Single or multiple target lesions measure ≥40 mm to ≤140 mm in overall length, with ≥60% diameter stenosis by operator's visual estimate.
* Patent popliteal artery (no stenosis ≥50%) distal to the treated segment.
* At least one patent infrapopliteal vessel (<50% stenosis) with run-off to the ankle.

Exclusion Criteria:

* Iliac stent in target limb that has required re-intervention within 12 months prior to index.
* Target vessel that has been treated with bypass surgery.
* PAD classified as Rutherford clinical category 0, 1, 5 or 6.
* Known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter or INR >1.8.
* Stroke diagnosis within 3 months prior to enrollment.
* History of unstable angina or myocardial infarction within 60 days prior to enrollment.
* Thrombolysis within 72 hours prior to the index procedure.
* Acute or chronic renal disease (e.g., as measured by a serum creatinine of >2.5 mg/dL or >220 umol/L), or on peritoneal or hemodialysis.
* Significant disease or obstruction (≥50%) of the inflow tract that has not been successfully treated at the time of the index procedure (success measured as ≤30% residual stenosis, without complication).
* No patent (≥50% stenosis) outflow vessel providing run-off to the ankle.
* Target lesion(s) requires percutaneous interventional treatment, beyond standard balloon angioplasty alone, prior to placement of the study stent.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2017-11-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Sullivan, MD, Principal Investigator — Minneapolis Heart Institute / Abbott Northwestern Hospital; Thomas Zeller, MD, Principal Investigator — Herz-Zentrum University Hospital; Masato Nakamura, MD, Principal Investigator — Toho University Ohashi Medical Center
Locations (43):
- United States (31):
  - Brookwood Medical Center, Birmingham, Alabama
  - Cardiology Associates of Mobile, Mobile, Alabama
  - Arizona Heart Hospital, Phoenix, Arizona
  - Yale New Haven Hospital, New Haven, Connecticut
  - Bradenton Cardiology Center, Bradenton, Florida
  - MediQuest Research Group/ Munroe Regional Medical Center, Ocala, Florida
  - Coastal Vascular, Pensacola, Florida
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Prairie Education and Research Cooperative, Springfield, Illinois
  - Kings Daughters Medical Center, Ashland, Kentucky
  - Endovascular Technologies / Grace Research, Bossier City, Louisiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Institute of the South, Lafayette, Louisiana
  - Michigan Outpatient Vascular Institute, Dearborn, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Michigan Vascular Center, Flint, Michigan
  - Minneapolis Heart, Minneapolis, Minnesota
  - Deborah Heart & Lung Center, Browns Mills, New Jersey
  - NC Heart & Vascular Research, Raleigh, North Carolina
  - WakeMed Research, Raleigh, North Carolina
  - Riverside Methodist Hospital, Columbus, Ohio
  - Doylestown Hospital, Doylestown, Pennsylvania
  - Pinnacle Health Harrisburg, Harrisburg, Pennsylvania
  - Berks Cardiologists, Wyomissing, Pennsylvania
  - North Central Heart, Sioux Falls, South Dakota
  - Kore Cardiovascular Research, Jackson, Tennessee
  - Austin Heart Research, Austin, Texas
  - Cardiovascular Specialist of TX / North Austin Medical Center, Austin, Texas
  - Grace Research, Huntsville, Texas
  - Mission Research Institute/Guadalupe Regional Medical Center, New Braunfels, Texas
  - Cardiovascular Associates of East Texas, Tyler, Texas
- Germany (6):
  - Karolinen-Hospital, Arnsberg
  - Universitaets-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - Westküstenklinikum Heide, Heide
  - Universitätsklinikum Leipzig AoR Leipzig, Leipzig
  - St. Bonifatius Hospital, Lingen
- Japan (6):
  - Kansai Rosai Hospital, Hyōgo
  - Kasukabe Chuo General Hospital, Kasukabe
  - Kokura Memorial Hospital, Kitakyushu-shi
  - Morinomiya Hospital, Osaka
  - Omihachiman Community Medical Center, Shiga
  - Toho University Ohashi Medical Center, Tokyo

REFERENCES:
- [Derived] Sullivan TM, Zeller T, Nakamura M, Gaines PA; MIMICS-2 Trial Investigators. Treatment of Femoropopliteal Lesions With the BioMimics 3D Vascular Stent System: Two-Year Results From the MIMICS-2 Trial. J Endovasc Ther. 2021 Apr;28(2):236-245. doi: 10.1177/1526602820980419. Epub 2020 Dec 17. PMID 33331207

RESULTS

PARTICIPANT FLOW:
Groups:
- BioMimics 3D Stent: Implantation of BioMimics 3D nitinol stent using the BioMimics 3D Stent System
Period: Overall Study
Arm/Group | BioMimics 3D Stent
Started | 271
30-Days Follow-up | 268
12-Months Follow-up | 256
24-Months Follow-up | 225
36 Months-Follow-up | 208
Completed | 208
Not Completed | 63
Not completed — Death | 24
Not completed — Lost to Follow-up | 18
Not completed — Withdrawal by Subject | 16
Not completed — Physician Decision | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 271
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91
  Male | 180
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 253
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 31
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 215
  More than one race | 0
  Unknown or Not Reported | 9

OUTCOME MEASURES:

1. Primary Outcome: Primary Safety Endpoint (Freedom From a Composite of Major Adverse Events (MAE)
Description: Freedom from a composite of major adverse events (MAE) comprising death, any major amputation performed on the target limb or clinically-driven target lesion revascularization (TLR) through 30 days.
Time Frame: 30 days
Population: Subjects with available 30 day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 269
Participants | 268

2. Primary Outcome: Primary Effectiveness Endpoint (Primary Stent Patency Rate)
Description: The primary effectiveness endpoint of the MIMICS-2 Study was defined as the primary stent patency rate at 12 months. Patency was defined as no significant reduction in luminal diameter (< 50% diameter stenosis) since the index procedure. Loss of patency was determined by an independent core laboratory when the peak systolic velocity ratio (PSVR) exceeds 2.0, or where angiography revealed > 50% diameter stenosis, or where the subject had a CDTLR.
Time Frame: 12 months
Population: Subjects were included in analysis population if they had imaging data qualifying as a 12m visit and/or subjects without imaging data who experienced a CDTLR through 12 months. Additionally, if a subject is missing stent patency status at the 12m window but found to be patent at a later out-of-window date, subject was considered patent at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 249
Participants | 182

3. Secondary Outcome: Secondary Safety (Overall MAE Rate at 30 Days)
Description: Contribution of individual MAE rates for death, major amputation performed on the target limb and clinically-driven target lesion revascularization to the overall MAE rate at 30 days.
Time Frame: 30 Days
Population: Subjects with available 30 day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 269
Participants
  Freedom from Death | 269
  Freedom from Major Amputation | 269
  Freedom from CD-TLR | 268

4. Secondary Outcome: Long Term Safety (Overall MAE Rate at Month 12)
Description: Overall MAE rate at Month 12 and contribution of individual event rates to the overall MAE.
Time Frame: 12 months
Population: Subjects are included in the analysis population if (i) they have sufficient follow-up (at least 12 months less 30 days), or (ii) they have had the event of interest (each event is considered separately).
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 261
Participants
  Freedom from MAE | 226
  Freedom from Death: number analyzed (Participants) | 260
  Freedom from Death | 257
  Freedom from Major Amputation: number analyzed (Participants) | 258
  Freedom from Major Amputation | 258
  Freedom from CD-TLR: number analyzed (Participants) | 259
  Freedom from CD-TLR | 227

5. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: Overall rate and incidence of type of serious adverse events from Day 0 through completion of Study follow-up at Month 36.
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 271
Participants
  total number of participants | 271
  All SAE (In-hospital) | 13
  All SAE (30 Days) | 26
  All SAE (12 Months) | 114
  All SAE (24 Months) | 146
  All SAE (36 Months) | 164

6. Secondary Outcome: Technical Success
Description: Percentage of subjects in which a final result of ≤50% residual diameter stenosis (in-stent) was achieved at index procedure
Time Frame: Procedural (at end of index procedure)
Population: Subjects with available baseline angiography
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 269
Participants | 269

7. Secondary Outcome: Primary Stent Patency
Description: Determined at Months-12 and 24 using values of: PSVR >2.0, >2.4; >2.5; and >3.5, each to indicate loss of patency on duplex ultrasound or where angiography reveals >50% diameter stenosis or where the subject undergoes clinically-driven TLR.
  Further analysis of the patency data purely using a reference PSVR of >2.4, >2.5 and >3.5 was not feasible from the data that was collected.
Time Frame: Months 12 & 24
Population: Relevant data was not collected to provide the outcome analysis
Groups:
- BioMimics 3D Stent: Implantation of BioMimics 3D nitinol stent using the BioMimics 3D Stent System
  BioMimics 3D Stent System: Femoropopliteal stenting
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Improvement of Rutherford Clinical Category by 1 or More
Description: Comparison of Rutherford Clinical Category measured at Baseline, Day 30, Months 12 and 24.
  Categories 0 - Asymptomatic
  1. - Mild claudication
  2. - Moderate claudication
  3. - Severe claudication
  4. - Ischemic rest pain
  5. - Minor tissue loss
  6. - Major tissue loss
Time Frame: Baseline, Day 30, Months 12 & 24
Population: Number of participants participating in the study changed at 30 Days, 12 Months and 24 Months
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 268
Participants
  Improvement of Rutherford Category of 1 or more at 30 Days | 233
  Improvement of Rutherford Category of 1 or more at 12 Months: number analyzed (Participants) | 254
  Improvement of Rutherford Category of 1 or more at 12 Months | 216
  Improvement of Rutherford Category of 1 or more at 24 Months: number analyzed (Participants) | 221
  Improvement of Rutherford Category of 1 or more at 24 Months | 195

9. Secondary Outcome: Clinical Outcome (Six-Minute Walk Test)
Description: Comparison of measured at Baseline, Day 30, Months 12 and 24 (subgroup of US investigational sites only).
Time Frame: Baseline, Day 30, Months 12 & 24
Population: Number of participants analysed changed over the time period
Measure: Mean (Standard Deviation); unit: yards
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 22
yards
  Baseline | 230 (162)
  30 Days: number analyzed (Participants) | 21
  30 Days | 349 (221)
  12 Months: number analyzed (Participants) | 15
  12 Months | 278 (143)
  24 Months: number analyzed (Participants) | 7
  24 Months | 405 (140)

10. Secondary Outcome: Functional Outcome (Ankle Brachial Index (ABI) Measurement)
Description: Comparison of the ankle brachial index (ABI) measurement at Baseline, within 30 days after index procedure, then at Months 12 and 24.
Time Frame: Baseline, Day 30, Months 12 & 24
Population: Number of participants assessed for ABI index measurement at Baseline, within 30 days after index procedure, then at Months 12 and 24.
Measure: Mean (Standard Deviation); unit: ABI
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 271
ABI
  ABI at Baseline: number analyzed (Participants) | 257
  ABI at Baseline | 0.70 (0.20)
  ABI at 30 Days: number analyzed (Participants) | 263
  ABI at 30 Days | 0.98 (0.16)
  ABI at 12 Months: number analyzed (Participants) | 247
  ABI at 12 Months | 0.92 (0.19)
  ABI at 24 Months: number analyzed (Participants) | 208
  ABI at 24 Months | 0.94 (0.20)

11. Secondary Outcome: Change of Walking Impairment Questionnaire Score
Description: Comparison of the Walking Impairment Questionnaire at Baseline, within 30 days after index procedure, then at Months 12 and 24.
  The WIQ consists of 3 primary categories assessing walking distance, stair-climbing, and walking speed, as previously described. Individuals are asked to rate the degree of difficulty of various activities with responses ranging from 0 (unable) to 4 (none).
Time Frame: Baseline, Day 30, Months 12 & 24
Population: Walking Impairment Questionnaire score at Baseline, within 30 days after index procedure, then at Months 12 and 24.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 270
scores on a scale
  Baseline WIQ score: number analyzed (Participants) | 266
  Baseline WIQ score | 0.28 (0.24)
  30 Days WIQ score: number analyzed (Participants) | 264
  30 Days WIQ score | 0.58 (0.32)
  12 Months WIQ score: number analyzed (Participants) | 253
  12 Months WIQ score | 0.58 (0.31)
  24 Months WIQ score: number analyzed (Participants) | 220
  24 Months WIQ score | 0.56 (0.31)

12. Secondary Outcome: Number of Participants With Freedom From Stent Fracture
Description: Stent integrity measured as freedom from fracture, defined as clear interruption of a stent strut observed in a minimum of two projections, determined by core lab examination of X-rays taken with the leg in extension at 12, 24 and 36 Months.
Time Frame: Months 12, 24 & 36
Population: Number of participants with no fracture in study stent at 12, 24 and 36 Months assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | BioMimics 3D Stent
Number analyzed (Participants) | 229
Participants
  Freedom from stent fracture at 12 Months | 229
  Freedom from stent fracture at 24 Months: number analyzed (Participants) | 204
  Freedom from stent fracture at 24 Months | 204
  Freedom from stent fracture at 36 Months: number analyzed (Participants) | 102
  Freedom from stent fracture at 36 Months | 102

ADVERSE EVENTS:
Time Frame: 36 months
Description: Site reported serious adverse events.
Arm/Group | BioMimics 3D Stent
All-Cause Mortality (participants affected / at risk) | 24/271
Serious Adverse Events (participants affected / at risk) | 164/271
Other Adverse Events (participants affected / at risk) | 177/271
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioMimics 3D Stent (N=271)
Restenosis of treated segment (Vascular disorders) | 47 (60)
Arterial stenosis (non-target) (Vascular disorders) | 38 (51)
Restenosis (Vascular disorders) | 14 (21)
Restenosis of treated vessel (Vascular disorders) | 12 (15)
Thrombosis (Vascular disorders) | 4 (4)
Limb ischemia (Vascular disorders) | 4 (6)
Dissection (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Pseudoaneurysm (Vascular disorders) | 2 (2)
Abrupt occlusion (Vascular disorders) | 1 (1)
Amputation (unplanned, spontaneous) (Vascular disorders) | 1 (1)
Aneurysm (Vascular disorders) | 2 (3)
Dissection (≥ Grade C) in target vessel requiring intervention (Vascular disorders) | 1 (1)
Embolization, distal (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Total occlusion of the peripheral artery (Vascular disorders) | 4 (6)
Angina (Cardiac disorders) | 10 (13)
Congestive heart failure (CHF) (Cardiac disorders) | 10 (14)
Atrial fibrillation (Cardiac disorders) | 10 (14)
Myocardial infarction (Cardiac disorders) | 13 (18)
Myocardial ischemia (Cardiac disorders) | 5 (6)
Cardiac arrhythmia (Cardiac disorders) | 4 (4)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Gastro-intestinal bleeding (Gastrointestinal disorders) | 3 (4)
Sepsis (Infections and infestations) | 6 (7)
Infected peripheral wound (Infections and infestations) | 1 (2)
Urinary tract infection (UTI) (Infections and infestations) | 3 (3)
Arterial occlusion/thrombus at puncture site (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complications (Injury, poisoning and procedural complications) | 2 (2)
Groin hematoma ≥ 5 cm, with or without surgical repair (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Stroke or other neurological complications (Nervous system disorders) | 5 (5)
Renal failure/renal insufficiency (Renal and urinary disorders) | 7 (7)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Allergic reaction (medication, contrast media, device, etc.) (Immune system disorders) | 1 (1)
Amputation (planned) (Vascular disorders) | 1 (1)
Bleeding from anticoagulant or antiplatelet medications s (Blood and lymphatic system disorders) | 1 (1)
Haemorrhage, with or without transfusion (Blood and lymphatic system disorders) | 1 (1)
Death (MAE if cardiovascular-related) (Cardiac disorders) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transient ischemic attack (TIA) (Nervous system disorders) | 1 (1)
Other (Investigations) | 95 (172)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BioMimics 3D Stent (N=271)
Angina (Cardiac disorders) | 18 (22)
Arterial stenosis (non-target) (Vascular disorders) | 50 (68)
Restenosis (Vascular disorders) | 18 (27)
Restenosis of treated segment (Vascular disorders) | 63 (77)
Restenosis of treated vessel (Vascular disorders) | 14 (18)
Vascular access complications (Injury, poisoning and procedural complications) | 14 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT02400905/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-25): https://cdn.clinicaltrials.gov/large-docs/05/NCT02400905/SAP_001.pdf